CLINICAL TRIAL: NCT05536596
Title: Pharmacological Treatment on the Recovery of Neurosensory Disturbance After Bilateral Sagittal Split Osteotomy: a Randomized, Double-blind Trial
Brief Title: Pharmacological Treatment on the Recovery of Neurosensory Disturbance After Bilateral Sagittal Split Osteotomy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Collaborators: Universidad de los Andes, Chile (Other)
Responsible Party: Principal Investigator, Pedro Sole Ventura, Principal Investigator, Surgeon, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PISV01
Record Dates: First submitted 2022-09-01; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Retrognathism; Prognathism; Orthognathic Surgery; Neurosensory Disorder
Keywords: Bilateral Sagittal Split Osteotomy; Neurosensory Disturbances
MeSH Terms: conditions — Retrognathia; Prognathism; Sensation Disorders | interventions — Orthognathic Surgery; Melatonin; Tablets; Hydroxocobalamin; Cytidine; Uridine

STUDY DESIGN:
Intervention Model Description: The participants will be assigned into 4 groups. Groups A, B and C will receive the medication (Melatonin, Hydroxycobalamin and combination UTP/CMP/hydroxycobalamin), whereas the Group P will receive placebo.
Who Masked: Participant, Care Provider
Masking Description: In order to maintain the blindness of subjects and the main surgeon, the drugs will be delivered in an identical brown non-translucent bag. The only one who will know about the assignament will be the second researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Citoneurone (Experimental): Groups A will receive the pharmacology treatment with 1.5 mg uridine triphosphate, 2.5 mg cytidine monophosphate and 1 mg hydroxycobalamin (Citoneurone). One capsule orally three times a day for 60 days as suggested by the manufacturer for patients with trauma - compressive peripheral neural disorders.
  Interventions: Procedure: Orthognathic Surgery; Drug: Centrum
- Melatonin (Experimental): Group B will receive the pharmacology treatment with 10 mg Melatonin. One capsule orally at night for 60 days.
  Interventions: Procedure: Orthognathic Surgery; Drug: Melatonin 10 MG Oral Tablet
- Hydroxycobalamin (Experimental): Group C will receive the pharmacology treatment with 1 mg hydroxycobalamin (vitamin B12). One capsule daily for 60 days.
  Interventions: Procedure: Orthognathic Surgery; Drug: Hydroxycobalamin
- Placebo (Placebo Comparator): The controls will receive 1 capsule placebo containing 5 mg starch to be taken once daily.
  Interventions: Procedure: Orthognathic Surgery

INTERVENTIONS:
Procedure: Orthognathic Surgery — Prognathism/Retrognathism correction through surgical procedures
  Other Names: Bilateral Sagittal Split Osteotomy
Drug: Melatonin 10 MG Oral Tablet — Group B will receive the pharmacology treatment with 10 mg Melatonin. One capsule orally at night for 60 days.
  Arms: Melatonin
Drug: Hydroxycobalamin — Group C will receive the pharmacology treatment with 1 mg hydroxycobalamin (vitamin B12). One capsule daily for 60 days.
  Arms: Hydroxycobalamin
Drug: Centrum — Groups A will receive the pharmacology treatment with 1.5 mg uridine triphosphate, 2.5 mg cytidine monophosphate and 1 mg hydroxycobalamin (Citoneuron). One capsule orally three times a day for 60 days as suggested by the manufacturer for patients with trauma - compressive peripheral neural disorders.
  Other Names: Citoneurone [Cytidine + Hydroxocobalamin, + Uridine]
  Arms: Citoneurone

SUMMARY:
The bilateral sagittal split osteotomy (BSSO) of the mandible is one of the most used surgical techniques to achieve a harmonious jaw relation in the context of orthognathic surgery. Nevertheless, one of its main complications is neurosensory damage to the inferior alveolar nerve, which can cause severe impact in the quality of life on patients who suffer from it permanently. The purpose of this randomized clinical trial is to provide rigorous scientific evidence of the pharmacological effect of 1) Melatonin, 2) combination uridine triphosphate (UTP), cytidine monophosphate (CMP), and hydroxycobalamin (UTP/CMP/hydroxycobalamin) and 3) hydroxycobalamin regarding neurosensory disturbances incidence and persistence after BSSO.

DETAILED DESCRIPTION:
The study will be done according to the international standards of the Helsinki convention for medical research and approved by the scientific ethics committee of Universidad de los Andes Clinic.

All subjects will give their signed consent to participate of this clinical research.

This clinical randomized trial will be double-blinded as both the patient and the surgeon will not know the treatment used until the experiment is over. The randomization will be done using "random.org" software to assign participants into 4 groups. Groups A, B and C will receive the medication, whereas the Group P will receive a placebo.

ELIGIBILITY:
Inclusion Criteria: Patients with dentomaxillofacial anomalies who present a complete mandibular dental arch and who have not undergone previous mandibular surgery.

Exclusion Criteria:

patients who:

* do not have sufficient information in their clinical records
* cannot be contacted
* do not attend their check-ups (for at least 24 postoperative months in cases with DNS)
* have refused consent to the use of their information for purposes of research.
* already undergoing Orthognathic Surgery
* with systemic conditions prone to alter recovery patterns or serious systemic diseases (decompensated metabolic disorders; neoplasms; osteodysplasias; neuropathies).
* pregnancy

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurosensory Activity | pre-operative
  Presence or absense of symptoms and signs such as hypoesthesia, pain, anesthesia, numbness, among others
Neurosensory Activity | 1 day postoperative
  Presence or absense of symptoms and signs such as hypoesthesia, pain, anesthesia, numbness, among others
Neurosensory Activity | 3 day postoperative
  Presence or absense of symptoms and signs such as hypoesthesia, pain, anesthesia, numbness, among others
Neurosensory Activity | 2 weeks postoperative.
  Presence or absense of symptoms and signs such as hypoesthesia, pain, anesthesia, numbness, among others
Neurosensory Activity | 1 month postoperative
  Presence or absense of symptoms and signs such as hypoesthesia, pain, anesthesia, numbness, among others
Neurosensory Activity | 2 month postoperative
  Presence or absense of symptoms and signs such as hypoesthesia, pain, anesthesia, numbness, among others
Neurosensory Activity | 6 month postoperative
  Presence or absense of symptoms and signs such as hypoesthesia, pain, anesthesia, numbness, among others
Neurosensory Activity | 12 month postoperative
  Presence or absense of symptoms and signs such as hypoesthesia, pain, anesthesia, numbness, among others
Neurosensory Activity | 18 month postoperative
  Presence or absense of symptoms and signs such as hypoesthesia, pain, anesthesia, numbness, among others

SECONDARY OUTCOMES:
Subjective Test | pre-operative, at day 1 and 3, at week 2, and at month 1, 2, 6, 12 and 18 after surgery.
  Subjective testing using a questionnaire and visual analogue scale. 0 = normal sensation, 10= more severe sensory deficit.
Objetive Test | pre-operative, at day 1 and 3, at week 2, and at month 1, 2, 6, 12 and 18 after surgery.
  The Semmes-Weinstein (SW) test of sensitivity to touch/pressure will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Sole, DMD, OMFS, Principal Investigator — Universidad de Los Andes

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available due to anonymity and ethical considerations.

REFERENCES:
- [Background] Alolayan AB, Leung YY. Resolution of neurosensory deficit after mandibular orthognathic surgery: A prospective longitudinal study. J Craniomaxillofac Surg. 2017 May;45(5):755-761. doi: 10.1016/j.jcms.2017.01.032. Epub 2017 Feb 12. PMID 28318920
- [Background] Teerijoki-Oksa T, Jaaskelainen SK, Forssell K, Forssell H, Vahatalo K, Tammisalo T, Virtanen A. Risk factors of nerve injury during mandibular sagittal split osteotomy. Int J Oral Maxillofac Surg. 2002 Feb;31(1):33-9. doi: 10.1054/ijom.2001.0157. PMID 11936397
- [Background] da Costa Senior O, Gemels B, Van der Cruyssen F, Agbaje JO, De Temmerman G, Shaheen E, Lambrichts I, Politis C. Long-term neurosensory disturbances after modified sagittal split osteotomy. Br J Oral Maxillofac Surg. 2020 Oct;58(8):986-991. doi: 10.1016/j.bjoms.2020.05.010. Epub 2020 Jul 4. PMID 32631751
- [Background] Seddon HJ. A Classification of Nerve Injuries. Br Med J. 1942 Aug 29;2(4260):237-9. doi: 10.1136/bmj.2.4260.237. No abstract available. PMID 20784403
- [Background] Schlund M, Grall P, Ferri J, Nicot R. Effect of modified bilateral sagittal split osteotomy on inferior alveolar nerve neurosensory disturbance. Br J Oral Maxillofac Surg. 2022 Oct;60(8):1086-1091. doi: 10.1016/j.bjoms.2022.04.001. Epub 2022 Apr 13. PMID 35606209
- [Background] Ylikontiola L, Kinnunen J, Oikarinen K. Factors affecting neurosensory disturbance after mandibular bilateral sagittal split osteotomy. J Oral Maxillofac Surg. 2000 Nov;58(11):1234-9; discussion 1239-40. doi: 10.1053/joms.2000.16621. PMID 11078134
- [Background] Yoshioka I, Tanaka T, Khanal A, Habu M, Kito S, Kodama M, Oda M, Wakasugi-Sato N, Matsumoto-Takeda S, Seta Y, Tominaga K, Sakoda S, Morimoto Y. Correlation of mandibular bone quality with neurosensory disturbance after sagittal split ramus osteotomy. Br J Oral Maxillofac Surg. 2011 Oct;49(7):552-6. doi: 10.1016/j.bjoms.2010.09.014. Epub 2010 Nov 10. PMID 21071118
- [Background] van Merkesteyn JP, Zweers A, Corputty JE. Neurosensory disturbances one year after bilateral sagittal split mandibular ramus osteotomy performed with separators. J Craniomaxillofac Surg. 2007 Jun-Jul;35(4-5):222-6. doi: 10.1016/j.jcms.2007.04.006. Epub 2007 Jul 30. PMID 17681774
- [Background] Colella G, Cannavale R, Vicidomini A, Lanza A. Neurosensory disturbance of the inferior alveolar nerve after bilateral sagittal split osteotomy: a systematic review. J Oral Maxillofac Surg. 2007 Sep;65(9):1707-15. doi: 10.1016/j.joms.2007.05.009. PMID 17719387
- [Background] Panula K, Finne K, Oikarinen K. Neurosensory deficits after bilateral sagittal split ramus osteotomy of the mandible--influence of soft tissue handling medial to the ascending ramus. Int J Oral Maxillofac Surg. 2004 Sep;33(6):543-8. doi: 10.1016/j.ijom.2003.11.005. PMID 15308252